CLINICAL TRIAL: NCT07121101
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase IIa Clinical Study to Evaluate the Safety, Efficacy and Kinetic Characteristics of TRD205 Tablets for Postoperative Analgesia After Unilateral Hip Arthroplasty
Brief Title: To Evaluate the Safety, Efficacy and Kinetic Characteristics of TRD205 Tablets for Postoperative Analgesia After Unilateral Hip Arthroplasty
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Collaborators: The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRD205-II-02
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Analgesia After Unilateral Hip Arthroplasty
Keywords: TRD205、postoperative analgesia after unilateral hip arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 200mg treatment group (Experimental): Administered orally every 12 hours for a total of four times；Take 400mg tablets for the first time and 200mg each for the other three times.
  Interventions: Drug: TRD205 tablets
- 400mg treatment group (Experimental): Administered orally every 12 hours for a total of four times；Take800mg tablets for the first time and 400mg each for the other three times.
  Interventions: Drug: TRD205 tablets
- 600mg treatment group (Experimental): Administered orally every 12 hours for a total of four times；Take 1200mg tablets for the first time and 600mg each for the other three times.
  Interventions: Drug: TRD205 tablets
- Placebo (Placebo Comparator): Administered orally every 12 hours for a total of four times；Take 6 tablets for the first time and 3 tablets each for the other three times
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: TRD205 tablets — Administered orally every 12 hours for a total of four times；Take TRD205 2 tablets and Placebo 4 tablets for the first time ，TRD205 1 tablets and Placebo 2 tablets each for the other three times
  Arms: 200mg treatment group
Drug: TRD205 tablets — Administered orally every 12 hours for a total of four times；Take TRD205 4 tablets and Placebo 2 tablets for the first time ，TRD205 2 tablets and Placebo 1 tablets each for the other three times.
  Arms: 400mg treatment group
Drug: TRD205 tablets — Administered orally every 12 hours for a total of four times；Take TRD205 6 tablets and Placebo 0 tablets for the first time ，TRD205 3 tablets and Placebo 0 tablets each for the other three times.
  Arms: 600mg treatment group
Drug: placebo — Administered orally every 12 hours for a total of four times；Take Placebo 6 tablets for the first time ，Placebo 3 tablets each for the other three times.
  Arms: Placebo

SUMMARY:
This is a phase IIa, multicenter ,randomized, double-blind, placebo-controlled study designed to evaluate the safety, efficacy and kinetic characteristics of TRD205 tablets for postoperative analgesia after unilateral hip arthroplasty

DETAILED DESCRIPTION:
This study used a placebo as a control to explore the safety, efficacy and pharmacokinetic characteristics of multiple administration of different doses of TRD205 tablets for postoperative analgesia after unilateral total hip replacement surgery

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the purpose and significance of this study, voluntarily participate in this study, voluntarily sign the informed consent form, and voluntarily comply with the trial procedures;
* 18 to 80 years of age, male or female;
* 18 kg/m 2 ≤ BMI ≤ 32 kg/m 2 , Incl. Cutoff ;
* American Society of Anesthesiologists (ASA) physical status I to II (Appendix 6);
* Unilateral total hip arthroplasty under general anesthesia is planned, and PCIA analgesia is expected to be required within 48 hours after surgery;
* Able to understand the study procedures and the use of various scales involved in this study, and able to communicate effectively with the investigators.

Exclusion Criteria:

* Known allergies or contraindications to the investigational drug and other drugs that may be used during the trial, and those who are not suitable for participating in the trial judged by the investigator;
* Use the following drugs within 5 half-lives before randomization (subject to the actual drug instructions, if the half-life is unknown, wash out according to 48h), including but not limited to: analgesic drugs (except specified in the protocol), anticonvulsants, sedative-hypnotic drugs (except used according to the protocol), anxiolytics, antidepressants, CYP3A4 enzyme inhibitors or inducers, etc., use of Chinese herbal medicine with clear analgesic effect assessed by the investigator within 7 days before randomization; sign the ICF to successfully use intra-articular injection of cocktail therapy (specific drugs include but not limited to local anesthetics such as ropivacaine, lidocaine, bupivacaine; analgesics such as morphine; steroid drugs such as dexamethasone and methylprednisolone); refer to the list of prohibited drugs for specific types;
* Patients who cannot take oral drugs after surgery as judged by the investigator;
* Combining the following:

  1. Patients who received ipsilateral hip surgery within 1 year before randomization;
  2. Patients who received hip surgery within 3 months before randomization;
  3. Patients scheduled for unilateral hip revision surgery;
  4. Patients who receive total hip arthroplasty due to developmental dysplasia of the hip Type III-IV (see Appendix 9 for Crowe classification), femoral or acetabular tumor, femoral neck fracture and/or femoral neck fracture (excluding old femoral neck fracture, which is treated with internal fixation removal + total hip arthroplasty), and are not suitable for this study at the investigator's discretion;
  5. Patients planning to undergo surgery at other sites at the same time during the study;
* Concomitant with other pain conditions that may confound the postoperative pain evaluation as judged by the investigator;
* Sitting systolic blood pressure ≤ 90 mmHg at screening, or sitting diastolic blood pressure ≤ 50 mmHg at screening, and clinically significant abnormalities as judged by the investigator;
* Heart rate < 50 beats/min or heart rate > 100 beats/min during the screening period, and clinically significant abnormalities as judged by the investigator; or QTcF > 450 ms in males and QTcF > 470 ms in females [calculated by Fridericia's formula: QTcF = QT/(RR0.33)]; or participants with a history of severe arrhythmia such as type II atrioventricular block or above, or a history of cardiac insufficiency;
* Patients complicated with severe liver, kidney, cardiovascular and cerebrovascular diseases, metabolic system diseases, and should not participate in this trial at the discretion of the investigator;
* Participants with malignant tumor who are not suitable for participating in the study as judged by the investigator;
* Patients complicated with mental system diseases (such as schizophrenia, depression, etc.), dementia, migraine, history of epilepsy, and unsuitable for participating in the trial judged by the investigator;
* History of psychotropic drug and narcotic drug abuse, drug abuse and alcoholism within 1 year before randomization, i.e., those who drink more than 2 units of alcohol on average per day (1 unit = 360 mL of beer or 45 mL of 40% liquor or 150 mL of wine);
* Abnormal blood routine at screening: neutrophil count < 1.5 × 10 9 /L; platelet count < 100 × 10 9 /L; hemoglobin (Hb) < 80 g/L;
* Abnormal liver function in the screening period: ALT and/or AST ≥ 1.5 times the upper limit of normal, or total bilirubin ≥ 1.5 times the upper limit of normal;
* Abnormal renal function in the screening period: serum creatinine (Cr) ≥ 1.5 times the upper limit of normal and/or dialysis participants;
* Abnormal coagulation function during screening period: prothrombin time (PT) prolonged by more than 3 seconds and/or activated partial thromboplastin time (APTT) prolonged by more than 10 seconds;
* Patients with positive syphilis antibody (Syphilis TP) and human immunodeficiency virus antibody (HIV-Ab) tests during the screening period who are not suitable for participating in the trial at the investigator's discretion;
* Pregnant or lactating women;
* Those who are unwilling or unable to take effective contraceptive measures during the study or 30 times after the study;
* Participated in other drug or device clinical study within 3 months before randomization (signed ICF and received the investigational drug/device or placebo treatment, for medication or treatment, start timing);
* Other conditions that the investigator considers inappropriate for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-26 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events | 5 days
  By evaluating security metrics such as AEs, SAEs and TEAEs to evaluate the safety of multiple administration of TRD205 tablets in patients with postoperative analgesia after unilateral hip arthroplasty.
The total dose of morphine was administered to the patient 0 to 48 hours after the operation | Within 48 hours after the first administration
  To evaluate the efficacy of multiple administration of TRD205 tablets in patients with postoperative analgesia after unilateral hip arthroplasty

SECONDARY OUTCOMES:
Peak Plasma Concentration（Cmax） | From 1 hour before the first administration to 48 hours after the last administration.
  To evaluate the pharmacokinetic (PK) of multiple administration of TRD205 tablets in patients with postoperative analgesia after unilateral hip arthroplasty
Minimum concentration （Cmin) | From 1 hour before the first administration to 48 hours after the last administration
  To evaluate the pharmacokinetic (PK) of multiple administration of TRD205 tablets in patients with postoperative analgesia after unilateral hip arthroplasty
Time to peak（Tmax） | From 1 hour before the first administration to 48 hours after the last administration
  To evaluate the pharmacokinetic (PK) of multiple administration of TRD205 tablets in patients with postoperative analgesia after unilateral hip arthroplasty
elimination half life（T1/2） | From 1 hour before the first administration to 48 hours after the last administration
  To evaluate the pharmacokinetic (PK) of multiple administration of TRD205 tablets in patients with postoperative analgesia after unilateral hip arthroplasty
Area under the plasma concentration versus time curve （AUC） | From 1 hour before the first administration to 48 hours after the last administration
  To evaluate the pharmacokinetic (PK) of multiple administration of TRD205 tablets in patients with postoperative analgesia after unilateral hip arthroplasty

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No